CLINICAL TRIAL: NCT05035862
Title: A Phase 1 Study to Evaluate Safety, Toxicity, and Potential Mechanisms of Interferon Gamma-primed Mesenchymal Stromal Cells (MSCs) for Moderate-to-severe Persistent Asthma
Brief Title: Mechanisms of Interferon Gamma-primed Mesenchymal Stromal Cells (MSCs) for Moderate-to-severe Persistent Asthma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study terminated due to funding ending.
Sponsor: Emory University (Other)
Collaborators: The Marcus Foundation (Other); Ossium Health, Inc. (Industry)
Responsible Party: Principal Investigator, Edwin Horwitz, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00002655; 2709 (Other Grant/Funding Number: The Marcus Foundation)
Record Dates: First submitted 2021-09-03; First posted 2021-09-05 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol; Interferon-gamma; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Infusion of γMSCs (Experimental): Escalating doses Dose escalation design with two dose levels. The low dose level involves a single intravenous infusion of γMSCs at 2x106 cells/kg. The high dose level involves a single intravenous infusion of γMSCs at 5x106 cells/kg.
  Interventions: Drug: Albuterol Sulfate; Drug: Interferon gamma-primed mesenchymal stromal cells (MSCs); Drug: Prednisone

INTERVENTIONS:
Drug: Albuterol Sulfate — Participants who experience symptoms of cough, dyspnea, chest tightness or wheezing will initiate use of albuterol (2 inhalations, 90 mcg/actuation) by metered dose inhaler (MDI) every 20 minutes for up to 1 hour and then every 4 hours if necessary.
Drug: Interferon gamma-primed mesenchymal stromal cells (MSCs) — IFNγ-primed bone marrow MSCs at a dose level of 2x106 cells/kg and a dose level of 5x106 cells/kg
  Other Names: Interferon gamma (IFNγ)-primed human bone marrow-derived mesenchymal stromal cells
Drug: Prednisone — Prednisone is recommended if the participant uses more than 12 inhalations of albuterol in 24 hours (excluding preventive use before exercise), or if the patient has ongoing symptoms for 48 hours or longer. The recommended prednisone dose for acute exacerbations is 2 mg/kg/day (maximum 60 mg) as a single dose for two days followed by 1 mg/kg/day (maximum 30 mg) as a single dose for two days. All administered doses will be rounded down to the nearest 10 mg.

SUMMARY:
This study is a two strata, dose escalation Phase I clinical trial designed to assess the safety and determine the maximal tolerated dose (MTD) of allogenic cord tissue derived MSCs (cMSCs, stratum 1) and allogeneic, interferon-γ primed bone marrow MSCs (γMSCs, stratum 2). Each stratum is designed to independently accrue 3 children at a dose level 1 of 2x106 cells/kg and 6 children at dose level 2 of 10x106 cells/kg, resulting in 9 children in each stratum. The primary objectives are to determine the safety and toxicity of allogeneic cord tissue derived MSCs and allogeneic interferon-γ primed bone marrow derived MSCs.

DETAILED DESCRIPTION:
Asthma affects one out of every 10 patients in the United States. Many of these patients have poor asthma symptom control. For example, patients with moderate-to-severe persistent asthma have ongoing symptoms and airway inflammation despite aggressive treatment with asthma medications. These patients are at increased risk for medication-related side effects and potentially life-threatening exacerbations. Novel therapies are critically needed for this population.

Mesenchymal stem cells (MSCs) are cells that reside in the bone marrow. MSCs are anti-inflammatory and also promote body tissue repair. This study will determine whether one form of MSCs called "interferon gamma-primed MSCs or γMSCs" are safe for patients with moderate-to-severe asthma.

Patients will receive a single intravenous infusion of γMSCs at either 2x10^6 cells/kg or 5x10^6 cells/kg. Up to 12 young adults will be enrolled. The total sample size will not exceed 24 participants.

The study will take place at Children's Healthcare of Atlanta (for patient activities) and at Emory University (for laboratory research activities). Participants will be identified from the asthma clinics at Children's Healthcare of Atlanta. Participants will complete up to 12 visits over 1 year and will be compensated for their time and travel. At the completion of the study, any samples remaining after experimentation will be de-identified and made available for future research.

While some study participants may receive no direct benefit from participating in this study, others may benefit from the close monitoring of their respiratory health, specialized asthma education, and general evaluation of their condition, including lung function tests. Some participants also achieve psychological benefit from participating in an important research study and from interaction with the study staff. It is also possible that the knowledge obtained from this study, such as identification of biomarkers, may assist in the creation of novel asthma therapies in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 30 years at the screening visit
* Physician diagnosis of asthma
* Onset of asthma during childhood
* Evidence of atopy, evidenced by allergic rhinitis, aeroallergen sensitization, elevated total immunoglobulin E (IgE) level based on age-dependent reference values, or blood eosinophil counts > or = 150 cells/microliter
* Moderate-to-severe persistent asthma as defined by the National Asthma Education and Prevention Program Expert Panel Report-4

Exclusion criteria at the screening visit include any of the following (*may be re-enrolled):

* A Panel Reactive Antibodies (PRA) test is positive for human leukocyte antigens (HLA) antibodies against the γMSC product
* Oral or injectable corticosteroid use within the two-week period prior to the screening visit.* Nasal corticosteroids may be used at any time during this trial at the discretion of the study's Medical Principal Investigator.
* Use of medications known to significantly interact with corticosteroid disposition within the two-week period prior to the screening visit, including but not limited to carbamazepine, erythromycin or other macrolide antibiotics, phenobarbital, phenytoin, rifampin, and ketoconazole*
* Presence of chronic or active lung disease other than asthma, including disorders of the airways or chest wall
* Current smoking or vaping
* History of premature birth before 35 weeks gestation
* Significant medical illness other than asthma, including thyroid disease, diabetes mellitus, sickle cell disease, Cushing's disease, Addison's disease, hepatic disease, immune deficiency, or concurrent medical problems that could require oral corticosteroids during the study or that would place the subject at increased risk of participating in the study
* A history of cataracts, glaucoma, or any other medical disorder associated with an adverse effect to corticosteroids
* History of adverse reactions to corticosteroids or short-acting bronchodilators or any of their ingredients
* Receiving allergen immunotherapy other than an established maintenance regimen (continuous regimen for ≥ 3 months)*
* Pregnancy or lactation
* If the participant is a female, failure to practice abstinence or use of an acceptable birth control method
* Inability to perform study procedures
* Current participation in another investigational drug trial
* Evidence that the participant may be unreliable or nonadherent, or may move from the clinical center area before trial completion

Exclusion criteria at the randomization/infusion visit include any of the following:

* Clinically significant deterioration in the level of asthma control, evidenced by:

  * Decrease in post-bronchodilator forced expiratory volume in one second (FEV1) of 15% (absolute change) compared to the post-bronchodilator FEV1 value obtained at the baseline visit, or
  * An asthma exacerbation
* Clinically significant thrombocytopenia, anemia, neutropenia or elevations in the white blood cell count, assessed at the screening visit
* Positive pregnancy test

The investigators will also ask participants to refrain from receiving new asthma therapies such as biologics until the final safety determination is made 7 days after the γMSC infusion (at study Day 14). They will also ask participants to refrain from participating in other interventional drug studies for the duration of their participation.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Change in number of adverse events and severe adverse events post-intervention | During the infusion, during the observation interval after the infusion (2 hours postinfusion), one day after the infusion, and at 7 to 30 days after the infusion (study day 14 to 37)
  This outcome will measure safety of allogeneic cord tissue derived MSCs and allogeneic interferon-γ primed bone marrow derived MSCs. Assessments will be made by physical examination and further investigation as indicated. Events will be classified according to the NIH Clinical Toxicity Criteria for Adverse Events (CTCAE), version 5. All recorded adverse events and serious adverse events will be documented and recorded. Their attribution to the γMSC product will be determined. Adverse events that may be attributable to the study product include dyspnea, cough, wheezing, respiratory failure, allergic reaction, anaphylaxis, and infusion-related reaction.
Number of grade ≥3 adverse reaction attributable to the γMSC product | 7 to 30 days post-infusion (study day 14 to 37)
  This outcome will measure toxicity. Toxicity is defined as any grade ≥3 adverse reaction and attributable to the γMSC product (attribution listed as at least probable), occurring from MSC infusion (at study day 7) through 7 days post-infusion (study day 14). Toxicity is considered unacceptable.

SECONDARY OUTCOMES:
Change in lung function test | Baseline, 7 to 30 days post-infusion (study day 14 to 37)
  Change in lung function test and asthma characterization will determine the clinical impact of MSC therapy
In- vivo trafficking of MSCs after intravenous infusion | 7 to 30 days post-infusion (study day 14 to 37)
  In vivo trafficking of MSCs after intravenous infusion
Upper airway inflammation of MSC treatment | 7 to 30 days post-infusion (study day 14 to 37)
  Upper airway inflammation will be determined by analysis of small molecule inflammatory constituents in exhaled breath condensate.
Circulating inflammatory cells of MSC treatment | 7 to 30 days post-infusion (study day 14 to 37)
  Circulating cell inflammation will be determined by flow cytometric analysis of peripheral blood cells and AbSeq analysis of peripheral blood cells.
Biophysical characteristics of the cell products and correlation with clinical outcome | 7 to 30 days post-infusion (study day 14 to 37)
  Characteristics of the γMSCs will be determined by comprehensive analysis at the Marcus Center for Therapeutic Cell Characterization and Manufacturing (MC3M)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Horwitz, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified participant data will be shared and will be made available
Supporting Information: Study Protocol
Time Frame: 12 months after publication of the primary outcome manuscript.
Access Criteria: Access will be limited to scientific investigators who wish to perform a secondary analysis of the data. These investigators must provide a written request and data analysis protocol for review by the Principal Investigator.